CLINICAL TRIAL: NCT03745833
Title: Medical Mindfulness: Virtual Reality Mindfulness Therapy for Anxiety and Pain Management in Adolescent and Young Adult Patients With Eating Disorders
Brief Title: Medical Mindfulness: Virtual Reality Mindfulness Therapy for Eating Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Megen Vo, Clinical Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 47146
Record Dates: First submitted 2018-11-13; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Eating Disorder; Anxiety; Abdominal Pain
MeSH Terms: conditions — Feeding and Eating Disorders; Anxiety Disorders; Abdominal Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will be shown a brief VR-based mindfulness intervention after meals.
  Interventions: Device: Virtual Reality Mindfulness

INTERVENTIONS:
Device: Virtual Reality Mindfulness — Participating patients will be provided with a VR headset (pre-programmed with mindfulness content) after lunch for 15 minutes with supervision while on strict bedrest. The headset will be collected following the intervention. Patients are currently provided with a post-meal survey following all meals as part of the standard of care, and will complete the survey following the lunchtime intervention.

SUMMARY:
Adolescents and young adults with eating disorders undergoing refeeding on an inpatient unit often experience abdominal pain and anxiety either as a result of their medical condition or as an expected side effect of nutritional rehabilitation. The purpose of this study is to assess if VR (Virtual Reality) mindfulness therapy is more or as effective as the standard of care (supportive care such as aromatherapy, heat packs, distraction, and nausea bands) for treating and/or preventing anxiety and pain in patients with eating disorders during the re-nourishment process. The anticipated primary outcome will be reduction of abdominal pain and anxiety with utilization of this intervention.

DETAILED DESCRIPTION:
In this study, investigators hope to 1) assess acceptance of VR mindfulness among inpatient adolescents and young adults with eating disorders 2) assess effects of VR mindfulness on perceived abdominal pain and 3) determine the impact of VR mindfulness on anxiety scores.

This study is designed to test the feasibility, acceptability and effectiveness of VR mindfulness in patients as they undergo various medical and nutritional therapies to treat their conditions.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the inpatient medical unit for refeeding for malnutrition

Exclusion Criteria:

* non-English speakers

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Abdominal pain | 1 hour after meals
  We will measure pre- and post-intervention pain scores using the validated Faces Pain Scale

SECONDARY OUTCOMES:
Anxiety | 1 hour after meals
  We will measure pre- and post-intervention anxiety scores using the validated Hamilton Anxiety Scale

IPD SHARING:
Plan to Share IPD: No